CLINICAL TRIAL: NCT02941406
Title: Reproducibility of Microperimetry Using Nidek MP3 (Microperimeter 3) in Healthy Subjects and Patients With Macular Disease - Pilot Study
Brief Title: MP3 (Microperimeter 3) Reproducibility in Healthy Subjects and Macular Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Vienna Institute for Research in Ocular Surgery (Other)
Responsible Party: Principal Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Principal Investigator, Vienna Institute for Research in Ocular Surgery
Other Study IDs: MP3_REP
Record Dates: First submitted 2016-10-17; First posted 2016-10-21 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-10

CONDITIONS: Macular Degeneration
Keywords: Retina; Perimetry
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy subjects: * Men and Women aged 18 and older
  * Normal findings in the medical history unless the investigator considers an abnormality to be clinically irrelevant
  * Normal ophthalmological findings unless the investigator considers an abnormality to be clinically irrelevant
- Age-related macular degeneration patients: * Men and Women aged 18 and older
  * Presence of a macular disease (such as dry or exudative age-related macular degeneration, diabetic maculopathy, epiretinal membrane)

SUMMARY:
The aim of the present study is to investigate the reproducibility of the MP3 and to compare the results with conventional perimetry using the Octopus 101 in healthy subjects and patients with macular disease.

ELIGIBILITY:
Inclusion criteria for healthy subjects

* Men and Women aged 18 and older
* Written informed consent
* Normal findings in the medical history unless the investigator considers an abnormality to be clinically irrelevant
* Normal ophthalmological findings unless the investigator considers an abnormality to be clinically irrelevant

Inclusion criteria for macular disease patients

* Men and Women aged 18 and older
* Written informed consent
* Presence of a macular disease (such as dry or exudative age-related macular degeneration, diabetic maculopathy, epiretinal membrane)

Any of the following will exclude a subject from the study:

* Any opacities (corneal scar, dense cataract) which interferes with the study relevant measurements
* Visual acuity < 0.1 (Snellen)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 10 healthy subjects 20 macular patients
Sampling Method: Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2015-07; Primary Completion 2016-01 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Reproducibility of retinal sensitivity measurements using microperimetry | Two measurement within one week
  Two study measurements are scheduled within one week. Test-retest reproducibility will be assessed for retinal sensitivity using the coefficient of repeatability and Bland-Altman diagrams.

SECONDARY OUTCOMES:
Comparison of reproducibility of retinal sensitivity measurements assessed with microperimetry and conventional perimetry | Two measurement within one week
  In addition to microperimetry conventional perimetry will be performed and reproducibility of both devices will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Findl, MD, Prof., Principal Investigator — Vienna Institute for Research in Ocular Surgery
Locations (1):
- Hanusch-Krankenhaus, Vienna, Vienna, Austria